CLINICAL TRIAL: NCT03756051
Title: Harms of Hepatocellular Carcinoma Surveillance in Patients With Cirrhosis
Brief Title: Harms of Hepatocellular Carcinoma Surveillance
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Parkland Health and Hospital System (Other); Baylor College of Medicine (Other); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Kaiser Permanente (Other)
Responsible Party: Principal Investigator, Amit Singal, Associate Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 102016-012; R01CA212008 (NIH)
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Physical Harms; Financial Harms; Overdiagnosis; Psychosocial Harms
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort: This study will collect prospective longitudinal data to characterize rates and identify correlates of a) physical harms due to follow-up tests, b) financial harms, and c) inappropriate screening using electronic medical record data and manual chart review. The study will also use surveys and semi-structured interviews to characterize rates and identify correlates of screening-related psychological harms, e.g. cancer specific worry, situational anxiety, mood disturbances, and decisional regret. Lastly, investigators will create and disseminate a balance sheet of benefits and harms to inform patients, providers, healthcare organizations, payers, and policymakers about the role of hepatocellular carcinoma screening in patients with cirrhosis.
  Interventions: Other: Prospective Longitudinal Data; Other: Surveys and Semi-structured Interviews

INTERVENTIONS:
Other: Prospective Longitudinal Data — We will prospectively follow the cohort using electronic medical record to document the hepatocellular carcinoma screening process and characterize physical and financial harms related to positive or indeterminate screening results and burden of inappropriate screening. Patients are anticipated to undergo hepatocellular carcinoma screening every 6-12 months, so each patient will have ~4-8 screening encounters over the study duration. We will use manual chart review to determine intent of ultrasound exams (screening vs. diagnostic) and test results. Receipt of follow-up tests after positive or indeterminate screening results will be identified through electronic medical record extraction using Current Procedural Terminology (CPT) codes for CT, MRI, and biopsy.
Other: Surveys and Semi-structured Interviews — We will use surveys and semi-structured interviews to characterize psychological harms after positive or indeterminate screening tests. Patient surveys will include patient-reported scales to measure psychosocial factors at three times points: baseline, 1 month after screening result, and 4 months after screening result. Semi-structured interviews will be conducted via telephone to explore patient attitudes toward risk perception, test follow-up, competing demands, and "downstream harms", particularly financial issues (e.g., out-of-pocket costs, access to insurance, and juggling hepatocellular carcinoma screening process completion with competing demands-work and family).

SUMMARY:
This study leverage a multi-center randomized controlled trial assessing screening-related benefits (i.e. early tumor detection, treatment eligibility, and overall survival) among a racially and socioeconomically diverse population of patients with cirrhosis. However, the randomized controlled trial was not budgeted to assess hepatocellular carcinoma screening-related harms. The goal of this study is to quantify physical, financial, and psychosocial harms across three healthcare settings.

DETAILED DESCRIPTION:
Leveraging a multi-center randomized controlled trial assessing screening benefits in a socioeconomically and racially diverse population of patients with cirrhosis followed in 3 healthcare settings over a 4-year period, this study aims to:

Aim 1: Assess the effect of hepatocellular carcinoma screening on a) physical harms due to follow-up tests, b) financial harms, and c) overdiagnosis in patients with severe liver dysfunction or comorbid illness, through electronic medical record data, manual chart review, and validated survey measures.

Aim 2: Assess the effect of hepatocellular carcinoma screening on screening-related psychosocial harms, e.g. cancer-specific worry, situational anxiety, mood disturbances, and decisional regret, through longitudinal validated measures and qualitative interviews.

Aim 3: Create and disseminate a balance sheet of benefits and harms to inform patients, providers, healthcare organizations, payers, and policymakers about the value of hepatocellular carcinoma screening in patients with cirrhosis.

Over a 4-year period, electronic medical record data will be used to compare screening-related physical and financial harms between patients undergoing and those not undergoing hepatocellular carcinoma screening. Psychosocial harms, as ascertained through longitudinal measurement of validated survey instruments and qualitative interviews, will be compared between patients with positive or indeterminate screening results and those with negative results or without any screening. Mixed-effect regression analysis will be used to determine if screening harms differed by factors at multiple levels including patient (e.g. degree of liver dysfunction), provider (e.g. subspecialty training), and healthcare organization (e.g. access to liver transplantation). This study will seamlessly complement data from the parent randomized controlled trial. By immediately translating these high quality data about hepatocellular carcinoma screening benefits and harms into a balance sheet, the investigators will facilitate patient-provider discussions, inform payer decisions about reimbursement, and guide policy decisions. These data are also crucial to identify modifiable and high-yield intervention targets and strategies to reduce hepatocellular carcinoma screening harms in the future.

ELIGIBILITY:
Inclusion and exclusion criteria of the parent randomized controlled trial are as follows:

Inclusion Criteria:

* Adult patients (≥ 21 years old)
* Cirrhosis
* Outpatient visit in year prior to randomization
* English or Spanish speaking

Exclusion Criteria:

* History of hepatocellular carcinoma
* History of liver transplantation
* Child Pugh C cirrhosis
* Significant comorbid conditions with life expectancy < 1 year, (e.g., extrahepatic malignancy)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from the parent randomized controlled trial will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 2871 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Physical Harms | 4 Years
  Physical harms (contrast injury, radiation exposure, and biopsy complications) can result from screening or follow-up testing and extends beyond medical complications to include discomfort. A binary outcome (harm vs. no harm) will be defined for each person and each type of physical harm (contrast injury, radiation exposure, biopsy, and any physical harm). We will report the point estimate and 95% confidence interval for the proportion of patients with each type of harm in each arm, stratified by health system. Using an intention-to-treat principle, we will use Chi squared test to compare the proportion of patients with physical harms between the screening and usual care arms, with a secondary analysis stratified by health system. We will also perform a sensitivity analysis based on test intent, in which we will only include tests (and corresponding harms) performed as a direct result of hepatocellular carcinoma screening.
Financial Harms | 4 Years
  Financial harms may include anticipated or real costs of hepatocellular carcinoma screening and diagnostic evaluation including, indirect costs such as missed work, and opportunity costs such as distraction from other health-related activities. Financial harms will be summarized for each arm using descriptive analyses as average and range of costs per person. Degree of financial harms will be compared between the hepatocellular carcinoma screening and usual care arms using Student T test, with a secondary analysis stratified by health system. In a secondary analysis, a mixed-effect model approach will be employed to identify patient-, provider- and system-level factors associated with financial harm.
Overdiagnosis | 4 Years
  Defined as hepatocellular carcinoma diagnoses that are unlikely to have an effect on mortality, specifically among patients with: 1) significant comorbid conditions or 2) severe liver dysfunction, i.e. Child Pugh C cirrhosis, who are not candidates for liver transplantation, at hepatocellular carcinoma diagnosis. For the primary analysis, Chi squared test will be used to compare the proportion of patients with overdiagnosis between the screening arm and usual care arm, stratified by health system.
Psychosocial Harms | 4 Years
  Patients will be divided into 4 categories: true positives, false positives, true negatives, and no screening. True positives will be defined as those who develop hepatocellular carcinoma within 6 months of the screening test; false positives as those who remain without hepatocellular carcinoma diagnosis during 6 months of follow-up; and true negatives as those with normal screening tests and without hepatocellular carcinoma diagnosis during 6 months of follow-up. Psychosocial harms (cancer-specific worry, situational anxiety, mood disturbances, and decisional regret) will be defined by change in survey scores from baseline and will be calculated at 1 month and 6 months for each patient.

SECONDARY OUTCOMES:
Patient-, Provider-, and System-level Factors Associated with Physical Harms | 4 Years
  As a secondary analysis, we will construct mixed-effect logistic regression models to identify patient-, provider-, and system-level factors associated with physical harms (contrast injury, radiation exposure, biopsy, and any physical harm). Models will include random effects for providers and health systems to account for potential correlation at different levels. Final models will include covariates identified by stepwise variable selection procedure and those considered clinically important a priori (BMI, race, liver dysfunction, and gastroenterology care). Statistical significance will be declared for p<0.05.
Patient-, Provider-, and System-level Factors Associated with Psychosocial Harms | 4 Years
  We will construct a mixed regression model with the outcome being decisional regret and covariates including patient-, provider- and system-level factors. Decisional regret score, ranging from 0 to 100, will be analyzed as a continuous outcome. The mixed model will include random effects for providers and systems to account for correlation at different levels. The model will include covariates identified through stepwise variable selection and those considered clinically important a priori (age, gender, race and ethnicity, liver dysfunction).
Physical Harms | 12 Months
  Physical harms (contrast injury, radiation exposure, and biopsy complications) can result from screening or follow-up testing and extends beyond medical complications to include discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Singal, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Singal AG, Daher D, Narasimman M, Yekkaluri S, Liu Y, Cerda V, Banala C, Khan A, Lee M, Seif El Dahan K, Murphy CC, Kramer JR, Hernaez R. Benefits and harms of hepatocellular carcinoma screening outreach in patients with cirrhosis: a multicenter randomized clinical trial. J Natl Cancer Inst. 2025 Feb 1;117(2):262-269. doi: 10.1093/jnci/djae228. PMID 39288308
- [Derived] Singal AG, Reddy S, Radadiya Aka Patel H, Villarreal D, Khan A, Liu Y, Cerda V, Rich NE, Murphy CC, Tiro JA, Kramer JR, Hernaez R. Multicenter Randomized Clinical Trial of a Mailed Outreach Strategy for Hepatocellular Carcinoma Surveillance. Clin Gastroenterol Hepatol. 2022 Dec;20(12):2818-2825.e1. doi: 10.1016/j.cgh.2021.12.014. Epub 2021 Dec 10. PMID 34902568